CLINICAL TRIAL: NCT05817604
Title: Stereotactic Body Radiotherapy (SBRT) for Medically Inoperable Localised Renal Tumors (SABINA Trial)
Acronym: SABINA
Status: Active, not recruiting | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Manuel Galdeano-Rubio, Radiation Oncologist, MD, MSc, Consorci Sanitari de Terrassa
Other Study IDs: SABINA
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Kidney Neoplasm; Renal Cancer; Inoperable Disease; SBRT; SABR
Keywords: Stereotactic Body Radiotherapy; Renal Cancer; Primary Localized Renal Cancer; Kidney Neoplasm; Radiotherapy; Inoperable Cancer; Stereotactic ablative radiotherapy; SBRT; SABR
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Localized Renal Cancer-One arm: Patients diagnosed with medically inoperable localized renal cancer [Size <7cm (cT1b)] based on TC, MRI or PET Image Study.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Tumors ≤ 4cm: Single SBRT 26Gy dose or Multifraction SBRT dose 14Gyx3 fraction-squeme.
  Tumors ≥ 4cm: Multifraction SBRT dose 14Gyx3 or 9Gyx5 fraction-squeme.

SUMMARY:
Study evaluating the activity and efficacy of Stereotactic Body Radiotherapy for the treatment of medically inoperable localized renal cancer

DETAILED DESCRIPTION:
Stereotactic Body Radiotherapy (SBRT) is a non-invasive alternative to surgery to control localized primary renal cell cancer (RCC) in medically inoperable patients. The kidney tumor has classically been considered radioresistant. Multiple retrospective series and few Phase II trial have studied the role of SBRT in localized renal tumors with favorable outcomes. Although large prospective studies are lacking, we evaluate the safety and effectiveness of SBRT for the treatment of renal cancer.

Participants will be allocated to recieve either single 26Gy fraction or Multifraction 3 - 5 fraction-squeme.

Assesment at regular intervals will estimate the activity and efficacy of the technique, evaluate tolerability, estimate survival, estimate distant failure rate, and renal function change after SABR.

Follow-up visits occur at 1month and every 3 months in the first year after SBRT, then every 6 months in the second year and then yearly until study closure.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of Renal tumor and/or highly suspected malignant neoplasm by CT, MRI or PET.
* Tumor Diameter >1cm - <7cm
* Tumor visible on CT planning
* Medically inoperable disease (or rejection of surgery)
* Karnofsky Index >70%
* >18 y.o.
* Informed Consent signature

Exclusion criteria:

* Non-oncological renal disease or autoinmunological disorder that does not recommend the treatment with radiotherapy.
* Previous local/regional RT
* Life expectancy <6 months
* Concomitance with other antineoplastic drugs

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with localized renal cancer selected by each tumor board from Consorci Sanitari de Terrassa (CST) collaborative group medical centers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Local relapse-free survival | Participants should be followed continuously during 5 years
  Local Control assessed by RECISTv1.1 criteria with TC, MRI or PET-scan

SECONDARY OUTCOMES:
Metastases-Free Survival | Participants should be followed continuously during 5 years
  Metastases-Free Survival assessed by RECISTv1.1 criteria with TC, MRI or PET-scan
Overall Survival | Participants should be followed continuously during 5 years
  Defined as the time from diagnose to the date of death from any cause.
Cancer Specific Survival | Participants should be followed continuously during 5 years
  Defined as the time from diagnose to the date of death from renal cancer.
Renal treatment-related adverse events | Participants should be followed continuously during 5 years
  Specific Renal Function-related adverse events measured by estimate Glomerular Filtration Rate
Non-Renal treatment-related adverse events | Participants should be followed continuously during 5 years
  Number of patients with Non-Renal treatment-related adverse events as assessed by Common Toxicity Criteria for Adverse Effects v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Galdeano-Rubio, MD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain